CLINICAL TRIAL: NCT00241449
Title: A Double-blind, Randomized, Multicentre Trial Comparing the Efficacy and Tolerability of 250mg of Faslodex (Long Acting ICI 182,780) With 20mg of Nolvadex (Tamoxifen) in Postmenopausal Women With Advanced Breast Cancer
Brief Title: A Trial Comparing the Efficacy and Tolerability of Faslodex With Nolvadex in Postmenopausal Women With Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9238IL/0025
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer; Metastasis
Keywords: Locally advanced breast cancer or metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Fulvestrant; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Tamoxifen
  Interventions: Drug: Tamoxifen
- 2 (Experimental): Fulvestrant
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — intramuscular injection 250 mg
  Other Names: Faslodex; ZD9238
  Arms: 2
Drug: Tamoxifen — 20 mg oral tablet
  Other Names: Nolvadex
  Arms: 1

SUMMARY:
The purpose of this study is to compare the efficacy of Faslodex (fulvestrant) to Nolvadex (tamoxifen) as first-line treatment for postmenopausal women with advanced breast cancer. Patients will be treated until disease progression or until the investigator has determined that treatment is not in the best interest of the patient, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmation of breast cancer. Evidence of breast cancer that is not considered amenable to curative treatment.

Postmenopausal women. Written informed consent to participate in the study.

Exclusion Criteria:

* Previous treatment with hormonal therapy unless that therapy was tamoxifen for adjuvant breast cancer. The use of tamoxifen must have ceased at least one year before this study.

Previous treatment with Faslodex. Any existing serious disease, illness, or condition that will prevent participation or compliance with the study procedures.

Treatment with an investigational or non-approved drug within one month of then start of the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 1998-11; Primary Completion 2007-03 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Time to disease progression (TTP) | At the time of data cut-off for this trial, the median overall duration of follow-up was 441 days, with a total of 434 (73.9%) randomised patients, including 47 patients from Japanese centres having progressed.
  It is considered that these results indicate that adequate data were available for obtaining clinically meaningful information for the primary efficacy endpoint of time to disease progression

SECONDARY OUTCOMES:
Objective response rate (ORR) | At the time of data cut-off for this trial, the median overall duration of follow-up was 441 days, with a total of 434 (73.9%) randomised patients, including 47 patients from Japanese centres having progressed.
  It is considered that these results indicate that adequate data were available for obtaining clinically meaningful information for the primary efficacy endpoint of time to disease progression
Duration of response (DoR) | At the time of data cut-off for this trial, the median overall duration of follow-up was 441 days, with a total of 434 (73.9%) randomised patients, including 47 patients from Japanese centres having progressed.
Time to treatment failure (TTF) | At the time of data cut-off for this trial, the median overall duration of follow-up was 441 days, with a total of 434 (73.9%) randomised patients, including 47 patients from Japanese centres having progressed.
Overall survival (OS) | At the time of data cut-off for this trial, the median overall duration of follow-up was 441 days, with a total of 434 (73.9%) randomised patients, including 47 patients from Japanese centres having progressed.
Quality of Life (QOL) and Tolerability. | At the time of data cut-off for this trial, the median overall duration of follow-up was 441 days, with a total of 434 (73.9%) randomised patients, including 47 patients from Japanese centres having progressed.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Oncology Medical Science Director, MD, Study Director — AstraZeneca
Locations (139):
- United States (24):
  - Research Site, Little Rock, Arkansas
  - Research Site, Fountain Valley, California
  - Research Site, La Jolla, California
  - Research Site, Orange, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Venice, Florida
  - Research Site, Decatur, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Mason City, Iowa
  - Research Site, Shreveport, Louisiana
  - Research Site, Gloucester, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Columbus, Ohio
  - Research Site, Meadowbrook, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Austin, Texas
  - Research Site, Galveston, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Temple, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Lacey, Washington
  - Research Site, Seattle, Washington
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, Rosario
- Australia (4):
  - Research Site, Camperdown
  - Research Site, Concord
  - Research Site, Heidelburg
  - Research Site, Melbourne
- Austria (2):
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (4):
  - Research Site, Antwerp
  - Research Site, Haine-Saint-Paul
  - Research Site, Hasselt
  - Research Site, Leuven
- Brazil (3):
  - Research Site, Belo Horizonte
  - Research Site, Goiânia
  - Research Site, São Paulo
- Canada (10):
  - Research Site, Edmonton, Alberta
  - Research Site, Penticton, British Columbia
  - Research Site, Saint John, New Brunswick
  - Research Site, Newmarket, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Weston, Ontario
  - Research Site, York, Ontario
  - Research Site, Chicoutimi
  - Research Site, Montreal
- Finland (3):
  - Research Site, Kotka
  - Research Site, Kuopio
  - Research Site, Rovaniemi
- France (8):
  - Research Site, Clermont-Ferrand
  - Research Site, Évreux
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Pierre-Bénite
  - Research Site, Rodez
  - Research Site, Rouen
  - Research Site, Tours
- Germany (3):
  - Research Site, Frankfurt
  - Research Site, Göttingen
  - Research Site, Rostock
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Pécs
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
- Research Site, Dublin, Ireland
- Israel (2):
  - Research Site, Ashkelon
  - Research Site, Haifa
- Italy (14):
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Forlì
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Reggio Calabria
  - Research Site, Reggio Emilia
  - Research Site, Rozzano
  - Research Site, Sassari
  - Research Site, Trieste
- Japan (13):
  - Research Site, Amagasaki
  - Research Site, Fukuoka
  - Research Site, Kitakyushu
  - Research Site, Kumamoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saitama
  - Research Site, Sapporo
  - Research Site, Suita
  - Research Site, Tokyo
- Mexico (2):
  - Research Site, Guadalajara
  - Research Site, Mexico City
- Research Site, The Hague, Netherlands
- New Zealand (2):
  - Research Site, Christchurch
  - Research Site, Palmerston North
- Poland (4):
  - Research Site, Bydgoszcz
  - Research Site, Krakow
  - Research Site, Szczecin
  - Research Site, Warsaw
- Research Site, Coimbra, Portugal
- Research Site, Moscow, Russia
- South Africa (3):
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Lyttelton Manor
- Spain (4):
  - Research Site, Badalona
  - Research Site, Guadalajara
  - Research Site, Madrid
  - Research Site, Málaga
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Research Site, Istanbul, Turkey (Türkiye)
- United Kingdom (18):
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Chelmsford
  - Research Site, Chorley
  - Research Site, Coventry
  - Research Site, Huddersfield
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Luton
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Northampton
  - Research Site, Nottingham
  - Research Site, Prescot
  - Research Site, Telford
  - Research Site, Whitehaven
  - Research Site, Worthing
  - Research Site, York